CLINICAL TRIAL: NCT02714673
Title: Management of Patients on Long Term Anticoagulation Therapy Undergoing a Primary Total Hip of Knee Replacement
Acronym: ADELC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association pour le Développement et l'Enseignement de la Chirurgie Réparatrice et Orthopédique (Other)
Responsible Party: Principal Investigator, Dr David BIAU, Associate Professor, Association pour le Développement et l'Enseignement de la Chirurgie Réparatrice et Orthopédique
Other Study IDs: ADECRO
Record Dates: First submitted 2016-03-07; First posted 2016-03-21 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ADELC: Cohort of patients on long term anticoagulation and undergoing a primary hip or knee replacement.
  Interventions: Drug: anticoagulation
- CONTROL: Cohort of patients not on long term anticoagulation and undergoing a primary hip or knee replacement.

INTERVENTIONS:
Drug: anticoagulation — anticoagulation refers to any long term effective anticoagulation including antivitamin K, direct oral anticoagulants. Aspirin, clopidogrel are not included
  Groups: ADELC

SUMMARY:
It is a multicenter, prospective, observational study of standard care. This study analyses the care of patients on long term effective anticoagulation therapy (ADELC) during a primary hip or knee arthroplasty.

The objectives of the study are to:

1. Identify clinical practices set up for patient care
2. Assess the type and the frequency of perioperative complications
3. Look for factors, related to patients or treatments, associated with the occurrence of these complications.

The main objective is to estimate the risks, adjusted and not, of postoperative complications associated to a long term anticoagulation by comparing patients under anticoagulation to a control group of patients having the same interventions but who are not under anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years
* Programmed for primary hip or knee arthroplasty.
* Effective dose of anticoagulant drugs intake for more than 1 month with the intention to resume it after the intervention for ADELC cohort; no effective dose of anticoagulant drugs intake for the control cohort.

Exclusion Criteria:

* Patient non opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on long term effective anticoagulation (ADELC) or not undergoing a primary hip or knee replacement
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-06-01; Primary Completion 2018-10-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
a composite criteria including the occurrence of one or more bleeding complications, major thrombotic events, or reoperation for any reason | up to 3 months

SECONDARY OUTCOMES:
The length of hospital stay | until end of study, an expected 12 months
  this is a continuous outcome measured. It measures the number of days from date of entry to the date of hospital discharge
The proportion of patients who are transfused during the hospitalization | up to day 15
The occurrence of a complication of grade 2 or more from Dindo and Clavien classification . | within 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Cochin, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: Undecided